CLINICAL TRIAL: NCT04201652
Title: Comparing Superficial vs. Deep Local Anesthetic Infiltration to Improve Patient Experience During Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, David Sauder, Orthopedic Surgery, Assistant Professor, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio 1439
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Carpal Tunnel; Carpal Tunnel Syndrome
Keywords: Local Anesthetic; WALANT
MeSH Terms: conditions — Median Neuropathy; Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two interventional groups for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superficial (Active Comparator): Intervention: Superficial local anesthetic infiltration.
  Interventions: Procedure: Superficial local anesthetic infiltration
- Deep (Active Comparator): Intervention: Superficial and deep local anesthetic infiltration.
  Interventions: Procedure: Deep local anesthetic infiltration

INTERVENTIONS:
Procedure: Superficial local anesthetic infiltration — Superficial infiltration of local anesthetic for carpal tunnel release.
  Arms: Superficial
Procedure: Deep local anesthetic infiltration — Deep and superficial infiltration of local anesthetic for carpal tunnel release.
  Arms: Deep

SUMMARY:
Hypothesis: When comparing superficial infiltration of local anesthetic to superficial and deep infiltration of local anesthetic in the setting of carpal tunnel release, the null hypothesis is that there will be no significant difference between the two techniques.

Background and study rationale: Carpal tunnel syndrome is a very common clinical problem with significant patient burden that can be reliably treated with surgical carpal tunnel release. To minimize operating room time burdens and to improve patient recovery time, this procedure is generally performed with the patient wide awake using local anesthetic. While the majority of patients are able to tolerate this type of procedure, there is always a possibility of some discomfort or pain experienced during the procedure. The investigators would like to compare two local anesthetic infiltration techniques to determine which is best to provide the least amount of pain or discomfort during a carpal tunnel release. The two methods are subcutaneous infiltration alone (superficial) and subcutaneous infiltration with infiltration into the carpal tunnel (deep).

Research Design: This study design is a prospective randomized control trial.

Methodology: Patients will be recruited and randomized on the morning of their surgery to undergo either superficial or superficial and deep local anesthetic infiltration using 10cc of 1% lidocaine with epinephrine buffered with 8.4% sodium bicarbonate. They will be blinded as to which group they are in.

Participants will complete the Boston Carpal Tunnel Questionnaire as a baseline for comparison as well as a brief questionnaire on demographics. After the procedure, participants will complete a short questionnaire about any pain experienced during the administration of the local anesthetic and during the procedure. Presence and intensity of pain during the procedure are the primary outcome of this study.

Secondary outcomes include pain rating at 2, 8, and 24 hours post-procedure and a follow up Boston Carpal Tunnel Questionnaire score at 3 months. The surgeon will also make note whether there is any visible evidence of damage to the median nerve from deep infiltration at the time of surgery.

Statistical Analysis: The two groups (superficial vs. deep) will be compared directly for each of the outcomes listed in the methodology.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Undergoing carpal tunnel release

Exclusion Criteria:

* Patients undergoing repeat carpal tunnel release
* Patients undergoing simultaneous procedures for other hand/wrist pathology at the time of carpal tunnel release (i.e. trigger finger release, Dupuytren's, etc.)
* Patients with a history of Rheumatoid Arthritis or a history or previous trauma or surgery to the local area (i.e. distal radius fracture)
* Patients who lack the capacity to provide informed consent or understand the nature of the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Intensity of Pain During Procedure: VAS | Immediately after the procedure
  Intensity of pain during the procedure, scored on a 10-point VAS (Visual Analogue Scale) for pain, where 0 is no pain and 10 is the worst pain possible.
Intensity of Pain During Local Anesthetic Infiltration: VAS | Immediately after the procedure
  Intensity of pain during the local anesthetic infiltration, scored on a 10-point VAS (Visual Analogue Scale) for pain, where 0 is no pain and 10 is the worst pain possible.

SECONDARY OUTCOMES:
Intensity of Pain Post-Procedure: VAS | 2, 8, and 24 hours after the procedure.
  Intensity of pain after the procedure, scored on a 10-point VAS (Visual Analogue Scale) for pain, where 0 is no pain and 10 is the worst pain possible.
Boston Carpal Tunnel Questionnaire Score | Before the procedure and 3 months after the procedure.
  Boston Carpal Tunnel Questionnaire Score. The minimum score is 19 and would indicate low symptom severity and the maximum score is 95 which would indicate high symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: David Sauder, MD, FRCSC, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iqbal HJ, Doorgakant A, Rehmatullah NNT, Ramavath AL, Pidikiti P, Lipscombe S. Pain and outcomes of carpal tunnel release under local anaesthetic with or without a tourniquet: a randomized controlled trial. J Hand Surg Eur Vol. 2018 Oct;43(8):808-812. doi: 10.1177/1753193418778999. Epub 2018 Jun 5. PMID 29871567
- [Background] Patil S, Ramakrishnan M, Stothard J. Local anaesthesia for carpal tunnel decompression: a comparison of two techniques. J Hand Surg Br. 2006 Dec;31(6):683-6. doi: 10.1016/j.jhsb.2006.08.008. PMID 17046117
- [Background] Pressman A, Doumit G, Rosaeg O, Bell M. A double-blind randomized controlled trial showing the analgesic and anesthetic properties of lidocaine E to be equivalent to those of ropivicaine and bupivacaine in carpal tunnel release surgery. Can J Plast Surg. 2005 Winter;13(4):173-6. doi: 10.1177/229255030501300401. PMID 24227926
- [Background] Lalonde D. Minimally invasive anesthesia in wide awake hand surgery. Hand Clin. 2014 Feb;30(1):1-6. doi: 10.1016/j.hcl.2013.08.015. Epub 2013 Nov 9. PMID 24286736
- [Background] Altissimi M, Mancini GB. Surgical release of the median nerve under local anaesthesia for carpal tunnel syndrome. J Hand Surg Br. 1988 Nov;13(4):395-6. doi: 10.1016/0266-7681_88_90163-5. PMID 3249135
- [Background] Tomlinson PJ, Field J. Warm or refrigerated local anaesthetic for open carpal tunnel release: a single blind randomized controlled study. J Hand Surg Eur Vol. 2010 Mar;35(3):232-3. doi: 10.1177/1753193409354138. Epub 2009 Dec 9. PMID 20007415
- [Background] Lee HJ, Cho YJ, Gong HS, Rhee SH, Park HS, Baek GH. The effect of buffered lidocaine in local anesthesia: a prospective, randomized, double-blind study. J Hand Surg Am. 2013 May;38(5):971-5. doi: 10.1016/j.jhsa.2013.02.016. Epub 2013 Apr 6. PMID 23566722